CLINICAL TRIAL: NCT04707547
Title: Immune Profile and Prognosis of Malignant Liver Tumors With Radiofrequency Ablation (RFA) Therapy
Acronym: RFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201812053
Record Dates: First submitted 2020-12-16; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Liver Cancer
Keywords: immune cells
MeSH Terms: conditions — Liver Neoplasms | interventions — Immunotherapy; Nivolumab; Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Radiofrequency Ablation (Experimental): Malignant Liver Tumors With Radiofrequency Ablation (RFA) Therapy
  Interventions: Procedure: Radiofrequency Ablation
- Radiofrequency Ablation combine with Nivolumab (Placebo Comparator): Malignant Liver Tumors With Radiofrequency Ablation (RFA) Therapy, and improving immune systems by Nivolumab
  Interventions: Biological: immunotherapy with Nivolumab

INTERVENTIONS:
Biological: immunotherapy with Nivolumab — After subjects had received radiofrequency ablation for two weeks, they were performed by immunotherapy with Nivolumab 200mg.
  Arms: Radiofrequency Ablation combine with Nivolumab
Procedure: Radiofrequency Ablation — The most commonly used local ablation is radiofrequency ablation. In this operation, a radio frequency probe is used to insert the liver cancer under ultrasound or computer tomography guidance, and then the radio frequency waves generated by the current oscillations locally heat the high temperature, causing the liver cancer cells to die.
  Arms: Radiofrequency Ablation

SUMMARY:
Clearing potential intrahepatic metastasis to prevent early recurrence after liver cancer treatment, there are no effective interventions so far. For secondary metastatic cancer, only the lesions visible under ultrasound can be used, one by one for local ablation and chemotherapy, but people may develop new tumor lesions. Therefore, the treatment of potential tumors and recurrent tumors after ablation is a very important clinical issue.

DETAILED DESCRIPTION:
Clearing potential intrahepatic metastasis to prevent early recurrence after liver cancer treatment, there are no effective interventions so far. For secondary metastatic cancer, only the lesions visible under ultrasound can be used, one by one for local ablation and chemotherapy, but people may develop new tumor lesions. Therefore, the treatment of potential tumors and recurrent tumors after ablation is a very important clinical issue. Therefore, this study will include primary liver cancer, as well as secondary metastatic malignant liver cancer, such as colorectal cancer, lung cancer, breast cancer, and other cancers with a high incidence in Chinese patients, and detection of immune cells by surgery, and through various biomarkers to explore its mechanism and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Disease characteristics: Patients with primary or metastatic liver cancer judged by histology
* Age: 20 years old or older
* Life expectation: at least 3 months
* Hematology:

  1. Platelet count: at least 50,000/mm^3
  2. Prothrombin time (PT) or partial thromboplastin time (PTT): no more than 1.5 times the control group
  3. Creatinine: no more than 2.5 mg/dl
* No pregnancy, no rhythm adjuster or other implantable device
* There are no uncontrollable responses to this study
* Other malignant tumors, except for therapeutic non-melanoma skin cancer or cervical cancer 5 years before entering the study inside.
* The number of liver tumors is less than three, the size is less than three centimeters, or the size of a single tumor is less than five centimeters, and those who want to undergo radiofrequency ablation are treated.
* The clotting time is normal and the number of platelets needs to be greater than 50,000, total bilirubin is less than 3 mg/dl, controllable ascites, no extrahepatic metastasis and portal vein invasion, and those who want to undergo radiofrequency ablation.
* The patient refuses or is unable to perform surgery (eg, If the age is too old, for those who want to undergo radiofrequency ablation).
* Patients and their families must fully understand and agree to perform radiofrequency ablation procedures.

Exclusion Criteria:

* There are people with central nervous system metastases.
* Measure lesions only by previous radiotherapy or topical treatment.
* Biliary obstruction did not undergo adequate drainage procedures prior to enrollment.
* White blood cells (WBC) are less than 3,500 / mm3 and absolute neutrophil count (ANC) is less than 1,500 / mm3, platelets less than 100,000 / mm3
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is greater than 5.0 times the upper limit of the normal range (ULN).
* Serum total bilirubin levels are equal to or greater than 2.0 mg / dl.
* Serum creatinine greater than 1.5 mg / dl.
* There are peripheral neuropathies greater than grade 1.
* Concomitant diseases that may accumulate via chemotherapy. For example, active, noncontrolled infection or other activity, non-control Systemic diseases such as congestive heart failure, angina pectoris, respiratory insufficiency, arrhythmia.
* Those who are treated concurrently with other research drugs or other anti-cancer therapies.
* Pregnant or lactating women, or women with fertility potential, unless reliable and appropriate methods of contraception are used.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Analysis of the number of CD8+ T | 6 weeks
  Analysis of the number of CD8+ T Using PBMC to analyze the number of CD8+ T that is NK, NKT, DC, and Monocyte. Four-time blood draws - 15 ml/each. Week 0- the data of CD8+T before RFA. Week 1- the data of CD8+T after RFA. Week 3- the data of CD8+T after participators received the vaccine which is Nivolumab 200mg in Week 2.
  Week 6- the data of CD8+T
  Compare with Week 0 and Week 1 data for analysis the difference of the ability of the immune system.
  Compare with Week 1 and Week 3 data, if week 3 data is higher than week 1, it means that immunotherapy with Nivolumab has effects to strengthen the immune system.
  Compare with Week 3 and Week 6 for analysis the effects of immunotherapy with Nivolumab have continued or not.
  Moreover, analyzed the difference in the immune system between participators who received the vaccine and no received vaccine from week 3 to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, PHD, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dromi SA, Walsh MP, Herby S, Traughber B, Xie J, Sharma KV, Sekhar KP, Luk A, Liewehr DJ, Dreher MR, Fry TJ, Wood BJ. Radiofrequency ablation induces antigen-presenting cell infiltration and amplification of weak tumor-induced immunity. Radiology. 2009 Apr;251(1):58-66. doi: 10.1148/radiol.2511072175. Epub 2009 Feb 27. PMID 19251937
- [Background] Cui J, Wang N, Zhao H, Jin H, Wang G, Niu C, Terunuma H, He H, Li W. Combination of radiofrequency ablation and sequential cellular immunotherapy improves progression-free survival for patients with hepatocellular carcinoma. Int J Cancer. 2014 Jan 15;134(2):342-51. doi: 10.1002/ijc.28372. Epub 2013 Aug 5. PMID 23825037
- [Background] Napoletano C, Taurino F, Biffoni M, De Majo A, Coscarella G, Bellati F, Rahimi H, Pauselli S, Pellicciotta I, Burchell JM, Gaspari LA, Ercoli L, Rossi P, Rughetti A. RFA strongly modulates the immune system and anti-tumor immune responses in metastatic liver patients. Int J Oncol. 2008 Feb;32(2):481-90. PMID 18202772
- [Background] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821